CLINICAL TRIAL: NCT00911313
Title: Letrozole Versus Combined Metformin and Clomiphene Citrate for Ovulation Induction in Clomiphene-Resistant Women With Polycystic Ovary Syndrome
Brief Title: Letrozole or Combined Metformin Clomiphene Citrate (CC) for Women With CC Resistant Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU- 059; FMH-012-G
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; clomiphene resistance; letrozole
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole; Metformin; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole tablets (Femara; Novartis Pharma, Switzerland)
- Metformin-CC (Active Comparator)
  Interventions: Drug: metformin HCl (Cidophage®; CID,Cairo, Egypt); Drug: CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt)

INTERVENTIONS:
Drug: Letrozole tablets (Femara; Novartis Pharma, Switzerland) — 2.5 mg letrozole daily from day 3 of the menses for 5 days
  Arms: Letrozole
Drug: metformin HCl (Cidophage®; CID,Cairo, Egypt) — metformin HCl 1500 daily for 6-8 weeks
  Arms: Metformin-CC
Drug: CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt) — 150 mg CC for 5 days starting from day 3 of menstruation
  Arms: Metformin-CC

SUMMARY:
The purpose of this study is to compare and determine the efficacy of letrozole administration to that of combined metformin and Clomiphene in infertile women with polycystic ovary syndrome (PCOS) not responding to treatment with Clomiphene alone.

DETAILED DESCRIPTION:
Withdrawal bleeding was achieved using 10 mg of dydrogesterone tablets for 10 days before stimulation. In the letrozole group, 2.5 mg of letrozole oral tablets (Femara; Novartis Pharma Services, Switzerland) daily from day 3 of the menses for 5 days, whereas all patients in the combined metformin-CC group) received metformin HCl [Cidophage®; Chemical Industries Development(CID), Cairo, Egypt], 500 mg three times daily for 6-8 weeks. Then after the end of this period, they received 150 mg CC (Clomid®; Global Napi Pharmaceuticals, Cairo, Egypt) for 5 days starting from day 3 of menstruation. Patients continued treatment for three successive cycles using the same protocol. Metformin was stopped only when pregnancy was documented.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing syndrome
* Androgen secreting tumors

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Principally the ovulation rate as well as the number of growing and mature follicles, serum E2 (pg/ml), serum P (ng/mL), and endometrial thickness (mm).

SECONDARY OUTCOMES:
The occurrence of pregnancy and miscarriage.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG, Principal Investigator — Mansoura University Hospital; Tarek Shokair, MD, Study Director — Mansoura University Hospital; Ahmed Badawy, MD.PhD., Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Holzer H, Casper R, Tulandi T. A new era in ovulation induction. Fertil Steril. 2006 Feb;85(2):277-84. doi: 10.1016/j.fertnstert.2005.05.078. PMID 16595197
- [Background] Siebert TI, Kruger TF, Steyn DW, Nosarka S. Is the addition of metformin efficacious in the treatment of clomiphene citrate-resistant patients with polycystic ovary syndrome? A structured literature review. Fertil Steril. 2006 Nov;86(5):1432-7. doi: 10.1016/j.fertnstert.2006.06.014. Epub 2006 Sep 27. PMID 17007847